CLINICAL TRIAL: NCT06833736
Title: Feasibility and Acceptability of a Digital Health App to Facilitate More Sustainable and Healthier Diets: Protocol for a Pilot Trial.
Brief Title: A Health App Using Recipes and Education Components to Facilitate Sustainable and Healthier Diets.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 28317; 204000 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-02

CONDITIONS: Nutrition; Sustainability; Mobile Health Technology (mHealth)
Keywords: Nutrition; Diet; Sustainability; Sustainable diets; Healthy eating; mHealth; Mobile apps; Behaviour change; Intervention; Recipe analysis; Acceptability; Feasibility; Randomised controlled trial; Pilot trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator)
  Interventions: Behavioral: General information
- Intervention group 1 (Experimental)
  Interventions: Device: The "See Yourself Differently" app
- Intervention group 2 (Experimental)
  Interventions: Device: The "See Yourself Differently" app + messages

INTERVENTIONS:
Device: The "See Yourself Differently" app — As the app has not been evaluated before in terms of its impact on dietary change, the first intervention group will have the app as it stands. The overall aim of the syd is to improve general wellbeing across several health-related domains, which is achieved through engaging with its main features (the daily plan, journal, user profile, and chat function).
  Arms: Intervention group 1
Device: The "See Yourself Differently" app + messages — The plant-forward recipes and information pages available on the app will be made more salient for app users in this group through sending them via targeted messages in the chat function at specific times. Each day, the information pages will be sent at 09:30 and the recipes will be sent at 13:00.
  Arms: Intervention group 2
Behavioral: General information — The (no app) control group will be sent general health and sustainability information via email immediately after randomisation is done. To incentivise participation in both baseline and follow-up assessments, the control group will be offered lifetime access to the app and a summary of their self-reported food intake at week 10. The control group will be sent one email reminder halfway through (week 5) to remind them that they are involved in the study, provide them with instructions on the follow-up assessment, and that they will receive the intervention and dietary feedback at week 10.
  Arms: Control group

SUMMARY:
This study is a pilot trial of a smartphone app to promote sustainable and healthy eating, running for 10 weeks. The app is called "See Yourself Differently" (syd), which aims to promote general wellbeing in the working population. The investigators are interested in the feasibility and acceptability of the plant-based recipes and information pages, so the focus will be on how people engage with these features and how they meet their needs.

Participants will be randomised into three groups:

1. General information (no app)
2. syd app (app as it stands)
3. syd app with recipes and food education messages (app + messages)

Data on demographics and food choice will be collected at the start and end of the intervention. A subset of participants will also take part in short interviews to talk about their experiences.

DETAILED DESCRIPTION:
Overall aim:

This pilot trial aims to understand the feasibility and acceptability of the syd app. The main focus is around the plant-based recipes and information pages delivered through the chat functionality.

Specific objectives:

The primary objective is to understand the feasibility and acceptability of setting up and running a trial with the syd app, focusing on the reach, adoption, implementation, and maintenance. The secondary objectives are to explore the indicative efficacy of the app in facilitating more sustainable and healthier diets, measured by a change in meat and legume intake, to what extent the recipes and information pages contribute to this effect, and whether there is a relationship between the self-perceived capabilities, opportunities and motivations to consume a sustainable and healthier diet.

Intervention:

The overall aim of syd is to enhance general wellbeing across nine domains, through completing activities and forming micro habits. The app has five main pages (Home, Daily Plan, Journal, Profile, and Chat). Users can input a goal, browse the 'activity pages', enter them into their daily plan, and complete them. When interacting with the app by completing activities, conversing in the chat, journaling or through other methods, the app calculates their 'life quality index' across all domains and presents this to users in the profile page. As the app focuses on multiple health behaviours rather than dietary change specifically, only some of the features are relevant to diet, mainly the 'activity pages' that contain food-related information and recipes. The information pages contain general information on certain aspects of diets for health and sustainability, quick tips in achieving dietary goals, and more detailed information on "What", "Why" and "How" one can adopt healthy dietary principles. The recipes are available for breakfast, lunch and dinner, and vary in their composition of healthy and sustainable foods. The chat function uses a large language model to converse and recommend content to users based on their engagement in the app overall, as well as the prompts users input into the chat.

Sample size:

The target sample size will be 99 (33 per arm), which will account for the possibility of 40% dropout in the first two weeks, which is typical for smartphone apps, and would still suffice the rule of thumb for 25 per group to be included in a pilot study to yield a small standardised effect size.

Outcomes:

Outcomes (and data) that will be collected and include 1) programme reach (population characteristics), 2) adoption of the app (participation and retention rates), 3) acceptability of the intervention (engagement with and usefulness of the app features), 4) implementation of delivering the intervention (compliance), 5) maintenance of the intervention (participant and organizational sustainability), and 6) efficacy of the intervention (indications of change in behavioural determinants and behaviours).

ELIGIBILITY:
Inclusion Criteria:

* Have a personal (not work) smartphone
* Have access to WiFi at home
* Have an out-of-home data package
* Be 18 years of age or older

Exclusion Criteria:

* Underweight for their age and gender
* Follow a restrictive diet (e.g., pregnant, breastfeeding, food intolerant/allergic, attempting to lose weight, diabetes, cardiovascular disease, or other long-term disease including eating disorders)
* Have a mental disability or learning difficulty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Adherence to intervention | From enrolment to the end of the intervention at 8 weeks
  Number of days participants log on to the app, measured using the app analytics

SECONDARY OUTCOMES:
Change in legume intake | Enrolment and at the end of the intervention at 8 weeks
  Self-reported dietary intake from two 24h dietary recalls, averaged into portions per day
Change in meat intake | Enrolment and at the end of the intervention at 8 weeks
  Self-reported dietary intake from two 24h dietary recalls, averaged into portions per day

CONTACTS AND LOCATIONS:
Locations (1):
- London School of Hygiene & Tropical Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to upload IPD and related data dictionaries available on LSHTM's data repository called Data Compass.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 10 years after the publication of results.
Access Criteria: The data will be provided to other researchers for use in secondary research upon reasonable request through LSHTM's Data Compass repository. The provision of data will be subject to information being provided on the research objectives and ethics status of the project. Ethical approval will need to be sought before receiving the data.